CLINICAL TRIAL: NCT03065803
Title: Clinical Assessment of Buccal Plate Expansion Technique Versus Guided Bone Regeneration Technique in Socket Preservation in The Esthetic Zone: A Randomized Controlled Clinical Trial
Brief Title: Buccal Plate Expansion Technique Versus Guided Bone Regeneration Technique in Socket Preservation in the Aesthetic Zone.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Passant Khaled Tayaa (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Passant Khaled Tayaa, Clinical professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dental socket preservation
Record Dates: First submitted 2017-02-11; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Bone Resorption After Tooth Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buccal plate expansion technique in dental socket preservation (Active Comparator): An internal osteotomy of the socket buccal plate will be performed with a piezotome (SurgyStar).
  Two vertical osteotomies and one horizontal osteotomy will be made to push the buccal plate outward from the socket. Two small cervical releasing incisions will be made in the mesiobuccal and distobuccal aspects of the socket to permit the displacement of the osteotomies in the area of keratinized tissue. The socket will be loaded with natural bovine bone mineral (cerabone). The biomaterial will be pressed to push the released buccal plate outward. A collagen bio absorbable membrane will be utilized to cover the socket. The collagen membrane plug will be stabilized on the top of the socket with a cross suture (silk 4/0).
  Interventions: Procedure: Buccal plate expansion technique for dental socket preservation
- Guided Bone regeneration technique for socket preservation (Other): On buccal side, two vertical incisions will be made at mesial and distal papilla of the adjoining teeth. These incisions will be stretched out past mucogingival junction. After full-thickness flap reflection on buccal and lingual sides, atraumatic tooth extraction utilizing periotome will be performed. The periosteum of buccal flap will be incised; this would permit coronal advancement of facial flap and a tension-free primary closure. Extraction sockets will be grafted with natural bovine bone mineral (cerabone). Collagen membrane will be trimmed and placed on the grafted socket and alveolar bone. Buccal and lingual/palatal flaps will be approximated utilizing interrupted simple loop and vertical mattress sutures (4/0) (Sadeghi et al., 2016).
  Interventions: Procedure: Guided bone regeneration technique for post-extraction dental socket preservation

INTERVENTIONS:
Procedure: Buccal plate expansion technique for dental socket preservation — An internal osteotomy of the socket buccal plate will be performed with a piezotome (SurgyStar).
  Two vertical osteotomies and one horizontal osteotomy will be made to push the buccal plate outward from the socket. Two small cervical releasing incisions will be made in the mesiobuccal and distobuccal aspects of the socket to permit the displacement of the osteotomies in the area of keratinized tissue. The socket will be loaded with natural bovine bone mineral (cerabone). The biomaterial will be pressed to push the released buccal plate outward. A collagen bio absorbable membrane will be utilized to cover the socket. The collagen membrane plug will be stabilized on the top of the socket with a cross suture (silk 4/0).
  Other Names: Internal corticotomy for buccal plate of bone in extraction socket for socket preservation
  Arms: Buccal plate expansion technique in dental socket preservation
Procedure: Guided bone regeneration technique for post-extraction dental socket preservation — After full-thickness flap reflection on buccal and lingual sides, atraumatic tooth extraction utilizing periotome will be performed.The periosteum of buccal flap will be incised; this would permit coronal advancement of facial flap and a tension-free primary closure. Extraction sockets will be grafted with natural bovine bone mineral (cerabone). Collagen membrane will be trimmed and placed on the grafted socket and alveolar bone.. Buccal and lingual/palatal flaps will be approximated utilizing interrupted simple loop and vertical mattress sutures (4/0)
  Arms: Guided Bone regeneration technique for socket preservation

SUMMARY:
Introduction and evaluation of a new technique for socket preservation involving internal expansion of the buccal plate of the extraction socket using internal flapless corticotomy and bone grafting the extraction socket with application of bioresorbable membrane biomaterials in comparison with the conventional guided bone regeneration technique for a conventional socket preservation method hoping to maintain or improve hard and soft tissue contour of the alveolar ridge post tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring tooth extraction in the maxillary anterior teeth and premolars ranging to the second premolar.
* Cause of tooth extraction is due to caries, trauma or failed endodontic treatment.
* Only teeth with intact buccal bone plate will be considered for this study.
* Patients who are cooperative, motivated and hygiene conscious.
* Patients whose age is >18 years

Exclusion Criteria:

* Systemic conditions/disease that contraindicated surgery.
* Patients on drugs that may compromise bone healing.
* Radiation therapy in the head and neck region or chemotherapy during the 12 months prior to surgery.
* Smokers.
* Patients with Psychologic disorder.
* Pregnancy or lactation.
* Presence of acute periodontal or periapical pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
measuring horizontal and vertical bone dimensions 4 months after the surgical intervention. | 4 months
  measuring the horizontal and vertical bone loss after socket preservation using cone beam computed tomography (CBCT).

IPD SHARING:
Plan to Share IPD: Yes
the data will be available for other scientists after the end of the study on www.clinicaltrials.gov , all data will be shared except patient contact or private data